CLINICAL TRIAL: NCT06458829
Title: Effects of an Implementation Program to Promote Atrial Fibrillation Screening in Primary Care Centers in China
Brief Title: Promoting Atrial Fibrillation Screening in Primary Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xi Cao, associated professor, Sun Yat-sen University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: Sunyatsenu
Record Dates: First submitted 2024-06-03; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation New Onset
Keywords: Atrial Fibrillation; Disease screening
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Stepped-Wedge Cluster Randomized Trial. Six community centers will be included. There will be three steps for intervention implementation. Tat each step, two centers will be randomly assigned to receive intervention, other centers will serve as control group or maintain post-intervention status.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive SEARCH-AF intervention which includes opportunistic screening and screening promoting strategies.
  Interventions: Behavioral: SEARCH-AF
- Control group (Active Comparator): All the control groups will finally receive the SEARCH-AF intervention.
  Interventions: Behavioral: SEARCH-AF

INTERVENTIONS:
Behavioral: SEARCH-AF — SEARCH-AF program will include opportunistic screening among old adults during primary care visits and promoting strategies. Promoting strategies will be developed based on the Consolidated Framework for Implementation Research framework which may include leadership engagement, policy support, providing screening resources, atrial fibrillation screening and management training. General practitioner or nurse in each health care center will implement point-on-care screening. The intervention will last for six months and followed up for another six months.

SUMMARY:
Atrial fibrillation is the most common sustained cardiac arrhythmia in adults. Due to the asymptomatic and paroxysmal nature (randomly and shortly occurring of atrial fibrillation, and can therefore remain unnoticed) of atrial fibrillation. Atrial fibrillation increases the risk of stroke five fold if left untreated.

Screening in old populations above age 65 years is helpful to find more atrial fibrillation cases. However, screening for atrial fibrillation is not well implemented in China. Thus, this project aims to promote atrial fibrillation screening in primary care centers in China. We will develop an intervention program (SEARCH-AF) and examine the effects (including the clinical effects and implementation effects) of program.

DETAILED DESCRIPTION:
Six health care centers in Guangzhou China will be included. We will adopt a stepped-wedge randomized trial design. Two health care centers will be randomly selected to receive the SEARCH-AF program at each step (a total of three steps).

The SEARCH-AF program will include opportunistic screening among those who aged 65 or above and screening promoting strategies. The A total of 4800 old adults will be screened for atrial fibrillation using a handheld single-lead ECG tool upon their visit to family doctor, with 800 for each health care center. The promoting strategy will be developed based on the Consolidated Framework for Implementation Research and include leadership engagement, policy support, providing screening resources, staff training on atrial fibrillation screening and management.

The whole study will last for 18 months. We will examine the intervention effects including clinical effects (atrial fibrillation detection rate, anticoagulation rate, atrial fibrillation related hospital visits, and stroke related end points) and implementation effects (cost-effectiveness of the intervention, compliance to atrial fibrillation screening ).

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years or above
* living in community

Exclusion Criteria:

* with a previous confirmed diagnosis of atrial fibrillation
* with implanted ICD or pacemaker
* unable to provide consent
* involving in other atrial fibrillation screening program

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 4800 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation detection rate | End of the intervention (T0), three-month (T1) and six-month (T2) after the intervention.
  Rate of newly detected atrial fibrillation. The data will be collected via medical records (primary care medical system) review and patient interview.

SECONDARY OUTCOMES:
Anticoagulation rate | Three-month and six-month post the intervention
  Anticoagulation rate among the newly detected atrial fibrillation cases. The data will be collected via medical records (primary care medical system) review and patient interview.
Cost-effectiveness | Six-month post the intervention
  Cost-effectiveness refers to the cost of screening for one atrial fibrillation and preventing for one stroke, respectively. It will be assessed using cost-effectiveness ratio. The cost of intervention will include the direct screening cost (screening tool, manpower for carrying out the screening, training on screening, leaflet etc), cost on anticoagulation (expense on oral anticoagulants) and stroke treatment (in-hospital and out-of-hospital cost on stroke treatment). The cost of control group will include the cost on anticoagulation(expense on oral anticoagulants) and stroke treatment (in-hospital and out-of-hospital cost on stroke treatment ). All the cost data will be collected using a patient-reported information sheet.
Atrial fibrillation associated events | Three-month and six-month post the intervention
  Including stroke, bleeding events associated with anticoagulation (referred to bleeding that requires in-hospital treatment), and death. The data will be collected via medical records (primary care medical system) and patient interview.
Atrial fibrillation related medical resource consumption | Three-month and six-month post the intervention
  Including the number of in-hospital and out-of-hospital visits due to atrial fibrillation. Such data will be collected using a patient-reported information sheet.
Compliance with atrial fibrillation screening | Three-month and six-month post the intervention
  Compliance with atrial fibrillation screening refers to the degree of general practitioner/nurse perform screening as requested during the follow-up. It will be calculated by the number of practitioners/nurses who remained in the screening during follow-up/ the initial number of practitioner/nurse performing the screening. Such data will be collected using a practitioner/nurse-reported information sheet.

CONTACTS AND LOCATIONS:
Overall Officials: Xi CAO, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No